CLINICAL TRIAL: NCT00827515
Title: A Phase 1, Randomized, Open-Label, Single Dose, 4-Way Crossover Study In Healthy Volunteers To Assess The Relative Bioavailability Of The Oral Powder In Capsule (PIC) And An Immediate Release (IR) Film-Coated Tablet Of PH-797804 In The Fed And Fasted State
Brief Title: Relative Bioavailability and Food Effect Study
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A6631025
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Pain
Keywords: Relative Bioavailability Effect of food
MeSH Terms: conditions — Pain | interventions — PH 797804

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- One (Experimental)
  Interventions: Drug: PH797804
- Two (Experimental)
  Interventions: Drug: PH797804
- Three (Experimental)
  Interventions: Drug: PH797804
- Four (Experimental)
  Interventions: Drug: PH797804

INTERVENTIONS:
Drug: PH797804 — Single oral dose of 5mg PH797804 as a powder in capsule formulation in the fasted state
  Arms: One
Drug: PH797804 — Single oral dose of 5mg PH797804 as a powder in capsule formulation in the fed state
  Arms: Two
Drug: PH797804 — Single oral dose of 5mg PH797804 as an immediate release tablet formulation in the fasted state
  Arms: Three
Drug: PH797804 — Single oral dose of 5mg PH797804 as an immediate release tablet formulation in the fed state
  Arms: Four

SUMMARY:
Initial studies have used a powder in capsule formulation of PH797804. In future studies an immediate release tablet will be used. The purpose of this study is to compare blood levels of PH797804 following an oral dose of the powder in capsule formulation and the tablet formulation. In addition the effect of food blood levels of PH797804 will be investigated

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects aged 21 to 55 years
* Healthy is defined as no clinical relevant abnormalities identified by a detailed medical history, full physical examination including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests
* Willing to use acceptable methods of contraception as outlined in the study protocol
* Body mass index between 18 to 30 kg/m2
* Subjects who are willing and able to comply with the scheduled visits, treatment plan and other study procedures

Exclusion Criteria:

* Subjects with evidence or history of clinically significant disease
* Pregnant or nursing females
* Females of childbearing potential who are unwilling or unable to use an acceptable method of nonhormonal contraception from at least 14 days prior to the first dose until day 15 of period 4
* Subjects with conditions possibly affecting drug absorption (eg gastrectomy)
* A positive approved immunoassay/ELISA blood test for TB
* Subjects with a history of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for men
* Subjects who have use prescription or nonprescription drugs, vitamins and/or dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication
* Subjects who have been administered medications capable of inducing hepatic enzyme metabolism (eg barbiturates, rifampin, carbamazepine, phenytoin or primidone) within 14 days (or 5 half-lives of the inducing agent, whichever is longer) of day 1 or within 28 days of administration of St John's wort

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-02; Primary Completion 2009-04 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Blood levels of PH797804 up to 336 hours after dosing in each treatment period | 336 hours

SECONDARY OUTCOMES:
Safety and tolerability of PH797804 in each treatment period up to 336 hours post-dose | 336 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6631025&StudyName=Relative%20bioavailability%20and%20food%20effect%20study%20